CLINICAL TRIAL: NCT00626873
Title: Microvascular Perfusion Sonographic Imaging to Detect Early Stage Ovarian Cancer
Brief Title: Contrast-Enhanced Ultrasonography in Diagnosing Early-Stage Ovarian Cancer in Patients With an Adnexal Mass Undergoing Surgery to Remove the Ovary
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Fishman, Professor Obstetrics, Gynecology and Reproductive Science, Director- Gynecologic Oncology Fellowship and National Ovarian Cancer Early Detection Program, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 09-0226; P30CA068485 (NIH); VU-VICC-GYN-0720; VU-VICC-061292; CDR0000584233
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2008-10

CONDITIONS: Ovarian Cancer
Keywords: ovarian germ cell tumor; ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Definity (Experimental): Definity - perflutren lipid microspheres, 1-10 microns in diameter, which is approved for the use in patients with suboptimal echocardiograms to opacify the left ventricular chamber and to improve the delineation of the left ventricular endocardial border, to enhance the visualization of the ovarian vascular system.
  Interventions: Drug: Definity; Other: medical chart review

INTERVENTIONS:
Drug: Definity — Definity - perflutren lipid microspheres, 1-10 microns in diameter, which is approved for the use in patients with suboptimal echocardiograms to opacify the left ventricular chamber and to improve the delineation of the left ventricular endocardial border, to enhance the visualization of the ovarian vascular system.
  Other Names: perflutren lipid microspheres
Other: medical chart review

SUMMARY:
RATIONALE: New diagnostic procedures, such as contrast-enhanced ultrasonography, may be an effective method of finding ovarian cancer.

PURPOSE: This clinical trial is studying how well contrast-enhanced ultrasonography works in diagnosing early-stage ovarian cancer in patients with an adnexal mass undergoing surgery to remove the ovary.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether use of a contrast agent improves the images of the ovaries during ultrasonography.

OUTLINE: This is a multicenter study.

Patients may undergo baseline transabdominal or transvaginal ultrasonography, if not already done. Patients then undergo contrast-enhanced transabdominal or transvaginal ultrasonography using perflutren lipid microspheres (Definity®) IV.

Pathology reports from tissue collected during subsequent oophorectomy is analyzed and compared with ultrasonography findings.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adnexal mass
* Scheduled to undergo surgical oophorectomy

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* No known respiratory failure as manifested by signs and symptoms of carbon dioxide retention or hypoxemia
* No pulmonary vasculitis
* No known history of severe emphysema
* No known history of pulmonary emboli
* No other condition that causes pulmonary hypertension due to compromised pulmonary arterial vasculature
* No known history of severe pulmonary hypertension (i.e., systolic pulmonary artery pressures > 90 mm Hg)
* No known history of congenital heart defect that creates a bidirectional or right-to-left shunt
* No worsening or clinically unstable congestive heart failure
* No known acute myocardial infarction or acute coronary syndromes
* No known serious ventricular arrhythmias
* Not at high risk for arrhythmia due to prolongation of the QT interval
* No known or suspected hypersensitivity to blood, blood products, or albumin
* No known hypersensitivity to perflutren
* No known or suspected hypersensitivity to octafluoropropane or any other ingredients of perflutren lipid microspheres (Definity®)
* No mental status problems, illiteracy, or other circumstance that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Ovarian microvascularity | 2 years
  To evaluate the use of contrast agents to depict the tumor microvascularity to detect ovarian cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur C. Fleischer, MD, Study Chair — Vanderbilt-Ingram Cancer Center; David Fishman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Result] Fleischer AC, Lyshchik A, Hirari M, Moore RD, Abramson RG, Fishman DA. Early detection of ovarian cancer with conventional and contrast-enhanced transvaginal sonography: recent advances and potential improvements. J Oncol. 2012;2012:302858. doi: 10.1155/2012/302858. Epub 2012 Apr 26. PMID 22619674